CLINICAL TRIAL: NCT04295512
Title: Adaptation and Implementation of an ASD Executive Functioning Intervention in Children's Mental Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Kelsey Dickson, Assistant Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS-2018-0147
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Mental Health Disorder; Executive Dysfunction
MeSH Terms: conditions — Autism Spectrum Disorder; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Community therapists delivering routine care to participant children with no training in Unstuck and on Target
- Unstuck and on Target Training (Experimental): Therapists enrolled in Unstuck and on Target Training
  Interventions: Behavioral: Unstuck and on Target

INTERVENTIONS:
Behavioral: Unstuck and on Target — Unstuck and on Target is a cognitive-behavioral treatment that directly addresses executive functioning and self-regulation deficits in ASD and ADHD. Unstuck and on Target is the first contextually-based executive functioning treatment that targets flexibility, goal-setting and planning through a cognitive behavioral program centered on self-regulatory scripts that are consistently modeled and reinforced. Unstuck and on Target will be adapted for use in mental health service settings. Mental health therapists will be trained in Unstuck and on Target and deliver to youth and caregivers.
  Arms: Unstuck and on Target Training

SUMMARY:
The purpose of this project is to conduct a feasibility test of an ASD executive functioning intervention adapted for mental health settings, including examining the effectiveness and process of implementing this adapted intervention in community mental health programs.

DETAILED DESCRIPTION:
This project will examine the implementation and effectiveness of an ASD executive functioning intervention, entitled Unstuck and On Target, adapted for use in community mental health clinics. Minimizing the impact of executive functioning deficits in youth has broad public health implications, including improving the effectiveness of mental health services for youth such as those with autism spectrum disorders (ASD) and attention-deficit/hyperactivity disorder (ADHD). Improved executive functioning also has the potential for improvement in real-world functioning, including daily living skills, mental health, and educational outcomes. Although Unstuck and On Target is an established evidence-based intervention, the effectiveness of this intervention in mental health settings has not been established. Therefore, the primary aim is to collect data on implementation outcomes of the adapted intervention, including feasibility, utility, and therapist fidelity, in mental health settings. The secondary aim is to collect data on the preliminary effectiveness of Unstuck and On Target adapted for mental health settings. This study has the potential to make a significant impact by building local capacity to serve school-age children with executive functioning deficits in routine service settings, and advancing the science on the effectiveness of an established evidence-based practice (Unstuck and On Target) for specific services settings. It will also produce generalizable knowledge about implementation that can be applied for this population/setting.

ELIGIBILITY:
Inclusion Criteria for Therapists:

1. Employed as staff or a trainee at participating clinic (publicly-funded mental health program)
2. Employed for at least the next 7 months (i.e., practicum or internship not ending in next 7 months).
3. Has an eligible client on current caseload (see below).

Inclusion Criteria for Child Participants

1. Child age 5-13 years.
2. Has a current ASD diagnosis on record.
3. English or Spanish speaking.

Exclusion Criteria for Child/ Parent Participants

1. Child does not present with executive functioning deficits.
2. Child does not meet criteria for ASD via case record, on the Autism Diagnostic Observation Scale or exhibit other clinical indicators of ASD

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Child and Adolescent Services Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickson KS, Aarons GA, Anthony LG, Kenworthy L, Crandal BR, Williams K, Brookman-Frazee L. Adaption and pilot implementation of an autism executive functioning intervention in children's mental health services: a mixed-methods study protocol. Pilot Feasibility Stud. 2020 Apr 27;6:55. doi: 10.1186/s40814-020-00593-2. eCollection 2020. PMID 32699642

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Numbers pertaining to those who started and completed don't match the protocol number. Participant numbers in fact exceeded the numbers for protocol enrollment with the exception of Usual Care: Children. Reason for this inconsistency is due to child recruitment at the start of the COVID 19 pandemic.
Groups:
- Usual Care: Therapist: Community therapists delivering routine care in a community health setting. Note: some therapists enrolled with more than one child.
- Unstuck and On Target Therapist: Community therapists trained in delivering Unstuck and On Target in a community health setting.
  Note: some therapists enrolled with more than one child.
- Usual Care: Children; Unstuck and On Target: Children: Children with suspected or diagnosed ASD receiving care with a participating therapist.
Period: Overall Study
Arm/Group | Usual Care: Therapist | Unstuck and On Target Therapist | Usual Care: Children | Unstuck and On Target: Children
Started (Started refers to provisionally enrolled participants. For therapists: consented to participate but did not enroll a child. For children: Family consented but child never completed cognitive assessment.) | 18 | 23 | 12 | 22
Completed (Completed refers to participants that consented and fully enrolled. For therapists: referred an eligible client and began implementation. For children: consented and underwent a cognitive assessment to begin implementation with participating therapist.) | 11 | 16 | 12 | 20
Not Completed | 7 | 7 | 0 | 2
Not completed — Lack of family response to schedule assessment | 0 | 0 | 0 | 2
Not completed — Therapist did not refer eligible family | 7 | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Numbers represent participating therapists and their yolked child participants. Note that some therapists participated with more than 1 child during the study.
  For 1 Usual Care: Therapist, partial baseline data is missing.
Groups:
- Usual Care: Therapists: Community therapists delivering routine care in a community health setting. Note: some therapists enrolled with more than one child.
- Unstuck and On Target: Therapists: Community therapists trained in delivering Unstuck and On Target in a community health setting. Note: some therapists enrolled with more than one child.
- Total: Total of all reporting groups
Arm/Group | Usual Care: Therapists | Unstuck and On Target: Therapists | Usual Care: Children | Unstuck and On Target: Children | Total
Number analyzed (Participants) | 11 | 16 | 12 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Total column represents the combined mean of therapist and child ages.
  years
    Age: number analyzed (Participants) | 10 | 16 | 12 | 20 | 58
    Age | 34.07 (8.1) | 35.69 (6.1) | 9.37 (2.37) | 9.43 (2.46) | 35.07 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Overall number represents child participants.
  Participants
    Sex: number analyzed (Participants) | 10 | 16 | 12 | 20 | 58
    Sex: Female | 9 | 14 | 2 | 8 | 33
    Sex: Male | 1 | 2 | 10 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall number represents child participants.
  Participants
    Ethnicity: number analyzed (Participants) | 10 | 16 | 12 | 20 | 58
    Ethnicity: Hispanic or Latino | 6 | 6 | 9 | 16 | 37
    Ethnicity: Not Hispanic or Latino | 4 | 10 | 3 | 4 | 21
    Ethnicity: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Overall number represents child participants. Population: Overall number represents child participants.
  Participants
    Race: number analyzed (Participants) | 10 | 16 | 12 | 20 | 58
    Race: American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
    Race: Asian | 2 | 2 | 3 | 0 | 7
    Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Race: Black or African American | 0 | 1 | 0 | 1 | 2
    Race: White | 6 | 10 | 6 | 11 | 33
    Race: More than one race | 2 | 2 | 3 | 7 | 14
    Race: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — All therapist and child participants reside in the Southwestern United States.
  Participants
    United States | 11 | 16 | 12 | 20 | 59
Child-Baseline Measures [Mean (Standard Deviation); unit: units on a scale] — The Social Responsiveness Scale measures social behavior differences associated with autism. Ratings from all subscales are summed to determine an overall score represented as T-scores (Mean=50, SD=10; Min=30; Max=95), with and higher scores reflecting more disruptive behaviors.
  The Wechsler Abbreviated Scale of Intelligence-2nd Edition is a standardized assessment of cognitive ability consisting of four subtests that yield a full score. Each score is represented as a standard score (Mean=100, SD=15; Min=40; Max=160), with higher scores reflective of higher functioning. Population: Baseline measures were only collected for enrolled children and not for therapists. Thus, therapist values are 0
  units on a scale
    Child- Social Responsiveness Scale, Baseline T Scores: number analyzed (Participants) | 0 | 0 | 12 | 20 | 32
    Child- Social Responsiveness Scale, Baseline T Scores |  |  | 74.17 (12.10) | 74.50 (9.81) | 74.37 (10.54)
    Child- Wechsler Abbreviated Scale of Intelligence 2nd Edition, Baseline Standard Scores: number analyzed (Participants) | 0 | 0 | 12 | 20 | 32
    Child- Wechsler Abbreviated Scale of Intelligence 2nd Edition, Baseline Standard Scores |  |  | 92.42 (13.42) | 83.63 (17.99) | 87.03 (16.71)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention Measure
Description: The Acceptability of Intervention Measure (AIM) measure includes four items assessing the acceptability of an intervention. Participants rate the intervention using a 5-point Likert scale (1- Completely Disagree to 5- Completely Agree), with a minimum score of 4 and maximum score of 20 and higher scores indicating higher acceptability. This measure were designed to assess mental health providers' perceptions regarding acceptability of an evidence-based intervention. This measure demonstrate good reliability and validity. Providers trained in Unstuck and On Target completed this measure. Scores are an overall mean score.
Time Frame: 6 months after starting implementation
Population: Measure only administered to Therapist intervention (Unstuck and On Target) group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapists- Unstuck and On Target: Community therapists trained and delivering Unstuck and On Target to participant children
Arm/Group | Therapists- Unstuck and On Target
Number analyzed (Participants) | 14
score on a scale | 4.58 (0.46)

2. Primary Outcome: Intervention Appropriateness Measure
Description: The Intervention Appropriateness Measure (IAM) measure includes four items assessing the appropriateness of an intervention. Participants rate the intervention using a 5-point Likert scale (1- Completely Disagree to 5- Completely Agree), with a minimum score of 4 and maximum score of 20 and higher scores indicating higher appropriateness. This measure was designed to assess mental health providers' perceptions regarding appropriateness of an evidence-based intervention. This measure demonstrate good reliability and validity. Providers trained in Unstuck and On Target completed this measure. Scores are an overall mean score.
Time Frame: 6 months after starting implementation
Population: Measure only administered to Therapist intervention (Unstuck and On Target) group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapists - Unstuck and On Target: Community therapists that received training and delivered Unstuck and On Target to child participants
Arm/Group | Therapists - Unstuck and On Target
Number analyzed (Participants) | 12
score on a scale | 4.62 (0.47)

3. Primary Outcome: Feasibility of Intervention Measure
Description: The Feasibility of Intervention Measure (FIM) measure includes 4 items assessing the feasibility of an intervention. Participants rate the intervention using a 5-point Likert scale (1- Completely Disagree to 5- Completely Agree), with a minimum score of 4 and maximum score of 20 and higher scores indicating higher feasibility. This measure was designed to assess mental health providers' perceptions regarding feasibility of an evidence-based intervention. This measure demonstrate good reliability and validity. Providers trained in Unstuck and On Target completed this measure. Scores are an overall mean score.
Time Frame: 6 months after starting implementation
Population: Measure only administered to Therapist intervention (Unstuck and On Target) group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapists- Unstuck and On Target: Community therapists trained to deliver Unstuck and On Target to child participants
Arm/Group | Therapists- Unstuck and On Target
Number analyzed (Participants) | 12
score on a scale | 4.5 (0.61)

4. Primary Outcome: Average of Provider Fidelity Throughout Implementation Period
Description: Provider adherence or fidelity to the Unstuck and On Target intervention will be measured through observational coding of provider in-session behaviors using the fidelity measure developed as part of the Unstuck and On Target intervention. Observers rate the provider's use of Unstuck and On Target on 9 components, using a 5-point (1 to 5) Likert scale, with higher scores indicating higher fidelity.
  For this report, a single, averaged value of all fidelity scores has been calculated per component.
Time Frame: A single, averaged value of all fidelity scores has been calculated. Average fidelity represents scores over the course of 6 months of therapist implementation. Table rows represent different aspects of fidelity that were scored.
Population: Community therapists randomized to either usual care or intervention condition working with youth clients with an autism spectrum disorder.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unstuck and On Target: Therapists randomized to receive training and deliver Unstuck and On Target
Arm/Group | Usual Care | Unstuck and On Target
Number analyzed (Participants) | 11 | 16
score on a scale
  Home Practice Review | 1.36 (0.56) | 3.26 (1.42)
  Content Delivery | 1.44 (0.84) | 4.74 (0.61)
  Use of Visuals | 2.10 (1.13) | 4.64 (0.66)
  Use of Handouts | 1.57 (0.82) | 4.70 (0.76)
  Use of Vocabulary | 1.75 (1.00) | 4.47 (0.67)
  Goal, Why, Plan, Do, Check | 1.25 (0.77) | 4.18 (1.05)
  Models Skills (Flexibility, planning) | 2.47 (0.78) | 3.95 (0.79)
  Use of More Positive Praise than Correction | 4.63 (0.44) | 4.79 (0.57)
  Use of Parent Engagement Strategies | 3.27 (1.37) | 4.00 (1.13)

5. Primary Outcome: Child Behavior Checklist
Description: Child Behavior Checklist (CBCL) is a parent-report measure of child problem behavior. The CBCL is divided into three broadband scales (Internalizing, Externalizing, and Total Problem Scores) and several associate subscale scores. For this study, only the broadband scales were utilized for analyses. Scores are represented as T-scores with a population mean of 50 with standard deviation of 10 and ranges from 30 (minimum) to 95 (maximum. Higher scores reflect more mental health symptoms. The values reported below represent the mean change in the T-scores from the Total, Internalizing, and Externalizing T-Scores from baseline to 6 months post intervention for each condition group. Negative values represent an overall decrease in symptoms (better outcome) while positive values representing an increase in problem behaviors (worse outcome) from baseline to post when looking at the condition groups as a whole.
Time Frame: At baseline and 6 months post-implementation.
Population: Children with suspected or diagnosed ASD receiving care with a participating therapist.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care: Children: Children with suspected or diagnosed ASD receiving care from a participating therapist.
- Unstuck and On Target: Children: Children with suspected or diagnosed ASD receiving care from a participating therapist trained in Unstuck and On Target.
Arm/Group | Usual Care: Children | Unstuck and On Target: Children
Number analyzed (Participants) | 12 | 20
units on a scale
  Change in Total Problem Score | -4.54 (6.22) | -2.33 (4.53)
  Change in Internalizing Behavior Score | -2.64 (6.38) | -1.67 (4.17)
  Change in Externalizing Behavior Score | -5.36 (5.35) | -1.87 (6.97)

6. Secondary Outcome: Eyberg Child Behavior Inventory
Description: The Eyberg Child Behavior Inventory is a 36 item questionnaire of child behavior. Caregivers of participating youth completed the questionnaire to assess their perceptions of their child's disruptive behaviors.
  The Eyberg Child Behavior Inventory Intensity Scale score measures the frequency of a child's behavioral problems and ranges from 36 (minimum value) to 352 (maximum). A score of 127 or higher is considered to be in the clinical range.
  The values reported below represent the mean change in the average T-score from baseline to 6 months post intervention for each condition group.
  Negative values represent an overall decrease in problem behaviors (better outcome) while positive values representing an increase in problem behaviors (worse outcome) from baseline to post when looking at the condition groups as a whole.
Time Frame: At baseline and 6 months post-implementation.
Population: Children with suspected or diagnosed ASD receiving care with a participating therapist.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Children- Usual Care: Children participating with therapists delivering usual care in a community health setting.
- Children- Unstuck and On Target: Children participating with therapists trained to deliver Unstuck and On Target in a community health setting.
Arm/Group | Children- Usual Care | Children- Unstuck and On Target
Number analyzed (Participants) | 12 | 20
units on a scale | -7.09 (8.47) | 1.85 (9.53)

7. Other Pre Specified Outcome: Wechsler Abbreviated Scale of Intelligence Second Edition- Block Design Subscale
Description: The Wechsler Abbreviated Scale of Intelligence Second Edition, is a brief measure of intelligence. We administered the Block Design subscale, a timed visual construction task that measures changes in nonverbal reasoning ability by assessing an individual's capacity to analyze and synthesize abstract visual stimuli, demonstrating visual-spatial skills, and coordinating visual perception with motor actions to replicate geometric patterns using colored blocks.The subtest is scored by converting the raw scores into scale scores using standardized norms. Scores range from 1 (minimum) to 19 (maximum) with an average of 10. Values below represent the change in subscale scaled scores from baseline to post-intervention for participating children. Negative values represent an overall decrease in nonverbal reasoning ability (worse outcome) while positive values represent and overall increase in nonverbal reasoning ability (better outcome).
Time Frame: At baseline and 6 months post-implementation.
Population: Children with suspected or diagnosed ASD receiving care with a participating therapist.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children- Usual Care | Children- Unstuck and On Target
Number analyzed (Participants) | 12 | 20
units on a scale | 5.18 (7.99) | .79 (6.29)

8. Other Pre Specified Outcome: Executive Functioning Challenge Task
Description: The Executive Functioning Challenge Task deliberately tests a child's ability to utilize key executive functions like planning and flexibility by presenting scenarios that reveal potential areas of difficulty in their executive functioning skills. The test yields Flexibility and Planning raw scores with a minimum of 0 and maximum of 8. Higher scores indicate greater impairment in executive functioning. A total executive functioning raw score is also calculated as the sum of planning and flexibility scores.
  Values below represent the change in average raw scores from baseline to post-intervention for participating children.
  Negative scores represent an overall decrease in executive functioning impairment (better outcome) while positive scores representing an increase in executive functioning impairment (worse outcome) from baseline to post when looking at the condition groups as a whole.
Time Frame: At baseline and 6 months post-implementation.
Population: Children with suspected or diagnosed ASD receiving care with a participating therapist.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children- Usual Care | Children- Unstuck and On Target
Number analyzed (Participants) | 12 | 20
units on a scale
  Change in Planning Score | -0.09 (1.81) | -2.21 (1.97)
  Change in Flexibility Score | -.82 (2.93) | -0.79 (1.63)
  Change in Executive Functioning Total Score | -.91 (4.01) | -3.00 (2.80)

9. Other Pre Specified Outcome: Behavior Rating Inventory of Executive Function Second Edition
Description: The Behavior Rating Inventory of Executive Function- Second Edition is a 63-item rating scale completed by caregivers to assess executive function impairment in children. T scores have a population mean of 50 and standard deviation of 10, with a minimum score of 30 and maximum score of 95. Scales assessed included the Behavioral Regulation Index, Emotion Regulation Index and Cognitive Regulation Index, together forming an overall composite score, the Global Executive Composite. Values below represent the change in T-scores scores from baseline to post-intervention for participating children. T scores at or above 70 are considered clinically significant.
  Scores represent the change in T scores from baseline to post. Negative values represent decrease in impairment (better outcome) while positive scores representing an increase in impairment (worse outcome) from baseline to post when looking at the condition groups as a whole.
Time Frame: At baseline and 6 months post-implementation.
Population: Children with suspected or diagnosed ASD receiving care with a participating therapist.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children- Usual Care | Children- Unstuck and On Target
Number analyzed (Participants) | 12 | 20
units on a scale
  Change in Behavioral Regulation Index T-Score | -2.82 (8.94) | -3.54 (5.39)
  Change in Emotion Regulation Index T-Score | -2.82 (10.42) | -0.31 (6.96)
  Change in Cognitive Regulation Index T-Score | -1.55 (7.09) | -2.62 (7.68)
  Change in Global Executive Composite T-Score | -2.82 (7.43) | -2.46 (6.12)

ADVERSE EVENTS:
Time Frame: Adverse events data monitored throughout the 2 year study. Broader oversight for adverse events was provided by a Data Safety and Monitoring Committee (DSMB) selected before data collection began. The DSMB met repeatedly during the study at an average of 2 times a year through study completion (average of 4 meetings over the 2 year duration of the study).
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Usual Care: Therapists: Community therapists delivering routine care to participant children with no training in Unstuck and on Target
- Unstuck and On Target: Therapists: Community therapists delivering Unstuck and On Target to participant children
Arm/Group | Usual Care: Therapists | Unstuck and On Target: Therapists | Usual Care: Children | Unstuck and On Target: Children
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/23 | 0/12 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/23 | 0/12 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/23 | 0/12 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care: Therapists (N=18) | Unstuck and On Target: Therapists (N=23) | Usual Care: Children (N=12) | Unstuck and On Target: Children (N=22)
No Adverse Events were observed during the course of the study (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — No Adverse Events were observed during the course of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT04295512/Prot_SAP_000.pdf